CLINICAL TRIAL: NCT00043043
Title: Rectal Abberant Crypt Foci And Other Intermediate Biomarkers For Sporadic Colorectal Neoplasia: Cross-Sectional Prevelance And Modulation By Celecoxib
Brief Title: Celecoxib in Preventing Cancer in Patients With Rectal Polyps or Colorectal Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000069498; NCI-02-C-0194; NCT00056615 (obsolete NCT alias)
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2004-11

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Celecoxib

INTERVENTIONS:
Drug: celecoxib

SUMMARY:
RATIONALE: Celecoxib may be effective in preventing colorectal cancer in patients who have a history of rectal polyps or colorectal neoplasia.

PURPOSE: Randomized phase II trial to study the effectiveness of celecoxib in preventing colorectal cancer in patients who have a history of rectal polyps or colorectal neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effects of celecoxib vs placebo on the number of rectal aberrant crypt foci in patients with premalignant rectal polyps or prior sporadic colorectal neoplasia.

Secondary

* Compare the effects of these drugs on proliferation index, apoptotic index, and gene expression patterns in ascending and descending colon tissue from these patients before and after treatment.
* Assess gene expression patterns in normal mucosa from the ascending vs descending colon in patients referred for screening, surveillance, or diagnostic colonoscopy.

OUTLINE: This is a randomized, double-blind, placebo-controlled, chemoprevention study. Patients are stratified according to age (18 to 49 vs 50 and over) and number of rectal aberrant crypt foci (5-9 vs 10 or more).

All patients undergo a baseline biomarker assessment and full colonoscopy to resect all neoplasms, quantitate rectal aberrant crypt foci, and biopsy rectal mucosa.

Depending on the results of the biomarker assessments, patients are randomized to 1 of 2 treatment arms. Patients with no adenomas of 5 mm or greater receive no further treatment.

* Arm I: Patients receive oral celecoxib twice daily.
* Arm II: Patients receive oral placebo twice daily. In both arms, treatment continues for 6 months in the absence of unacceptable toxicity.

All patients undergo an endoscopic exam of the colorectum at completion of study.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for the baseline biomarker assessment and a total of 40 patients (20 per arm) will be accrued for the chemoprevention study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Age 18 to 49 with one of the following colorectal abnormalities:

  * At least one adenoma that is at least 1 cm
  * At least 3 adenomas of any size with at least 5 rectal aberrant crypt foci (ACFs)
* Age 50 and over with one of the following colorectal abnormalities:

  * At least one adenoma that is at least 5 mm and at least 5 rectal ACFs
  * History of polyps (at least 1 adenoma) within the past 5 years
* No history of germline cancer syndrome
* No stage III or IV colorectal cancer (Dukes' C or D) diagnosed within the past 6 months
* No current colorectal cancer
* No inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)

PATIENT CHARACTERISTICS:

Age

* See Disease Characteristics
* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin greater than 11.5 g/dL
* WBC greater than 3,000/mm^3
* Platelet count greater than 125,000/mm^3
* No significant bleeding disorder

Hepatic

* AST and ALT no greater than 1.5 times upper limit of normal (ULN)
* Bilirubin no greater than 1.5 times ULN
* Alkaline phosphatase no greater than 1.5 times ULN
* No chronic or acute hepatic disorder

Renal

* Creatinine no greater than 1.5 times ULN
* No chronic or acute renal disorder

Cardiovascular

* No uncontrolled hypertension
* No unstable angina
* No congestive heart failure

Pulmonary

* No asthma
* No severe chronic obstructive pulmonary disease

Gastrointestinal

* No active gastrointestinal ulcers
* No history of peptic ulcer disease

Other

* No prior hypersensitivity reaction to NSAIDs, aspirin, or sulfa drugs
* No medical contraindication to NSAID use
* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use effective contraception
* No known allergic reaction to indigo carmine
* No other clinically significant medical condition or abnormal laboratory value that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Anticipated use of corticosteroids less than 2 weeks over 6 months
* Anticipated use of mometasone less than 4 weeks over 6 months

  * No other concurrent inhaled steroids for 30 days before or during study participation

Radiotherapy

* No prior pelvic radiotherapy

Surgery

* Not specified

Other

* More than 30 days since prior investigational drugs
* No prior participation in this study
* No regular nonsteroidal anti-inflammatory drug (NSAID) or aspirin use (average of 3 or more doses per week for at least 3 months) except low-dose aspirin for cardiovascular disease prophylaxis
* No other concurrent investigational drugs
* No concurrent fluconazole or lithium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Hawk, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Naval Medical Center, Bethesda, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland